CLINICAL TRIAL: NCT07086859
Title: Alveolar Ridge Preservation Using Autogenous Whole Tooth Graft With 1 %Metformin :A Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Hassan Gadallah, Masters Degree Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 279
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dimensional Changes After Tooth Extraction; Tooth Extraaction; Socket Preservation
Keywords: Alveolar ridge preservation; socket preservation; Autogenous Whole tooth Graft; AWTG; Tooth grafting; tooth extraction; bone graft

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant
Masking Description: The patients participating in this clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test (Experimental): Autogenous Whole tooth graft + Metformin in the socket of extracted non-molar tooth
  Interventions: Procedure: TEST 1
- Control (Active Comparator): Autogenous whole tooth graft
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: TEST 1 — Autogenous whole tooth graft with metformin
  Arms: Test
Procedure: Control — Autogenous whole tooth graft
  Arms: Control

SUMMARY:
This study describes a technique used to preserve the bone dimensions after the tooth extraction inorder to facilitate later on the dental implant placement

DETAILED DESCRIPTION:
Socket preservation by type of graft used from the tooth combined with Metformin to enhace the results of the bone formation

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* patients requiring single extraction of non-molar tooth
* extraction sockets having more than 50% buccal alveolar bone loss

Exclusion Criteria:

* Pregnancy
* smokers
* patients not maintaing good oral hygiene
* presernce of acute endodontic infection in the tooth to be ectracted
* medical conditions hindering implant placement
* uncontrolled diabetes
* Immune suppression
* bisphosphanates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic buccolingual width ridge loss | 6 months
  Measuring the CBCT these dimensions pre operative and after 6 months

SECONDARY OUTCOMES:
Alveolar buccal ridge height, lingual ridge height | 6 months
  Measuring them on CBCT pre operative and after 6 months
the area percentage of newly formed bone, soft tissue and residual graft | 6 months
  By Histology after taking a biopsy after 6 months
Patient satisfaction evaluation | 2 weeks
  by visual analog scale (0-10)
Total number of analgesics taken in the first week | 1 week
  by asking the patient
Socket wound healing score | 2 weeks
  by taking occlusal clinical pictures of socket

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univeristy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elfana A, El-Kholy S, Saleh HA, Fawzy El-Sayed K. Alveolar ridge preservation using autogenous whole-tooth versus demineralized dentin grafts: A randomized controlled clinical trial. Clin Oral Implants Res. 2021 May;32(5):539-548. doi: 10.1111/clr.13722. Epub 2021 Mar 1. PMID 33565656
- See also: Related Info — https://doi.org/10.21608/ajdsm.2021.66398.1181
- See also: Related Info — https://doi.org/10.1097/SCS.0000000000004263